CLINICAL TRIAL: NCT00536744
Title: Use of the dermaPACE™ (Pulsed Acoustic Cellular Expression) Device in Conjunction With Standard of Care in the Treatment of Diabetic Foot Ulcers
Brief Title: Effectiveness of dermaPACE™ Device and Standard Treatment Compared to Standard Treatment Alone for Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SANUWAVE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAN07-DERM01
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active PACE application - 4 applications (Active Comparator): Application of acoustical pulse energy (extracorporeal shockwaves) to target ulcer + standard of care
  Interventions: Device: acoustical pulse energy (extracorporeal shockwave)
- Inactive, non-energy application (Sham Comparator): Non-energized (inactive - Sham)) application + standard of care
  Interventions: Other: Sham

INTERVENTIONS:
Device: acoustical pulse energy (extracorporeal shockwave) — Acoustical pulse energy (extracorporeal shockwave) + Standard of care wound dressing.
  Other Names: dermaPACE
  Arms: Active PACE application - 4 applications
Other: Sham — Non-energized (inactive - Sham) application + standard of care
  Arms: Inactive, non-energy application

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the dermaPACE Device to sham application, when administered in conjunction with standard treatments used in the treatment of DFUs.

DETAILED DESCRIPTION:
The objective of this clinical study is to compare the safety and effectiveness of the dermaPACE (Pulsed Acoustic Cellular Expression) Device to sham application, when administered in conjunction with the standard of care, in the treatment of DFUs.

Diabetic patients are susceptible to chronic foot ulcerations due to the effects of the diabetic's systemic disease halting the wound healing process. In the United States, 20.8 million people with active diabetes, and 41 million with pre-diabetic symptoms account for $132 billion dollars in healthcare costs per year. In 2002, 82,000 non-traumatic lower-limb amputations were performed on diabetics, corresponding to 60% of all lower limb amputations, usually preceded by a non-healing foot ulceration. Given the magnitude of this disease and the long-term effects and morbidity of amputation, DFUs require immediate and aggressive treatment to ascertain the best possible outcome for the diabetic patient.

Despite the development of advanced wound care products, there is still a need to find the most effective treatment for reducing the time required to close a DFU. At any given time, 3-4% of diabetics (600,000 patients) have a foot ulcer, and $2.5 billion was spent in 2002 in the United States treating DFUs. The average cost for a single episode of a foot ulcer has been reported to be $4,595.00 to $28,691.00. Shock wave devices, which utilize acoustic pressure waves, have been used for about 30 years in urology for lithotripsy. In the last decade this technology has gained FDA approval to treat chronic plantar fasciitis and lateral epicondylitis conditions that do not respond to conservative treatments (OssaTron® SANUWAVE, manufacturer). Further, clinical reports have indicated efficacy in treating many other orthopedic conditions including pseudoarthroses, calcification of the joints and avascular necrosis. This technology has also been shown to promote healing in several wound-healing applications, and it is worthwhile to continue to seek the full potential of this technology in wound healing.

Acoustic pressure waves initiate a biological response at the cellular level-stimulating production of angiogenic growth factors, including endothelial nitric oxide synthase (ENOS), vascular endothelial growth factor (VEGF), and proliferating cell nuclear antigen (PCNA). These factors are important components of the normal wound healing process. This cellular activation and growth factor expression stimulated by acoustic pressure wave treatment could play a decisive role in overcoming cell quiescence and increasing growth factor titers to levels sufficient to overcome proteases. This leads to the in-growing of newly formed vessels, and the increased cellular proliferation and tissue regeneration needed to heal a wound.

Clinical publications have recently reported the pressure wave induced mechanism described above can initiate and accelerate healing in burns, traumatic wounds and reconstructive skin flaps, and diabetic wounds. A pilot study using the dermaPACE device, performed in nine diabetic subjects with chronic leg ulcers has shown that this technology in patients with a history of chronic ulcers may achieve wound closure. Treatment with dermaPACE has the added benefits of being non-invasive and devoid of significant clinical side effects. Therefore, the objective of this study is to examine the safety and effectiveness of the dermaPACE acoustic pressure wave treatment device in combination with standard of care for the treatment of foot ulcers in diabetic patients.

The dermaPACE should offer an improved non-invasive standard of care that may shorten an otherwise lengthy healing process and therefore make later operative measures unnecessary. Given that conservative therapy may not be effective, dermaPACE may become a preferable alternative that would carry minimal risk based on the expected clinical outcomes described in this protocol. dermaPACE may improve patient quality of life when conservative therapy is not effective as well as provide a cost savings for the health care system.

ELIGIBILITY:
Major Inclusion Criteria:

* Male or female ≥ 18 years of age
* Diabetes mellitus
* One or more chronic foot ulcers (only one will be treated) that are located in the ankle area or below that has persisted a minimum of 30 days prior to the Screening visit
* HbA1c ≤ 12%
* Diabetic Foot Ulcers ≥ 1 cm2 and ≤ 16 cm2
* Ulcer Grade I or II, Stage A according to the University of Texas Diabetic Wound Classification system
* Ankle Brachial Index (ABI) ≥ 0.7 and ≤ 1.2, OR toe pressure > 50 mmHg, OR tcPO2> 40 mmHg.

Major Exclusion Criteria:

* Subject is morbidly obese (Body Mass Index ≥ 40)
* Subjects on dialysis
* Diagnosis of foot ulcer involving osteomyelitis
* Has evidence of prior ulcer in the same area
* Multiple diabetic foot ulcers on the foot that either are connected by fistulas or are within 5 cm of the target ulcer
* Subject's foot ulcer intended for study application has decreased in volume by 50% or more at the end of the two-week Run-in period as compared to the Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jorgensen, MD, Study Director — SANUWAVE, Inc.
Locations (23):
- United States (21):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - HOPE Research Insititute, Phoenix, Arizona
  - Southern Arizona VA Healthcare System (SAVAHCS), Tucson, Arizona
  - Center for Clinical Research, Castro Valley, California
  - Veterans Administration Long Beach Healthcare, Long Beach, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Fairfield County Foot Surgeons, Norwalk, Connecticut
  - Emory Orthopedic and Spine Center, Atlanta, Georgia
  - Northwestern Univ. Div. of Plastic Surgery, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Center for Palliative Wound Care; Calvary Hospital, The Bronx, New York
  - St. Vincent's Charity Hospital, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Nashville Family Footcare, Nashville, Tennessee
  - Richard Galperin, DPM, PA, Dallas, Texas
  - Complete Family Foot Care, McAllen, Texas
  - Robert Wunderlich, DPM, PA, San Antonio, Texas
  - Aurora Health Care, Milwaukee, Wisconsin
- Mathias Spital, Rheine, Germany
- Kings College Hospital, London, United Kingdom

REFERENCES:
- See also: Company Web Site — http://www.sanuwave.com

RESULTS

PARTICIPANT FLOW:
Groups:
- dermaPACE Application + Standard of Care: dermaPACE application + standard of care
  dermaPACE: dermaPACE + Standard of care wound dressing.
- Non-energized (Inactive) Application + Standard of Care: Non-energized (inactive) application + standard of care
  Sham: Sham treatment + Standard of care wound dressing.
Period: Overall Study
Arm/Group | dermaPACE Application + Standard of Care | Non-energized (Inactive) Application + Standard of Care
Started | 107 | 99
Completed | 78 | 71
Not Completed | 29 | 28
Not completed — Adverse Event | 13 | 10
Not completed — Death | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 7 | 8
Not completed — PI tried alternative treatment | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- dermaPACE Application + Standard of Care: dermaPACE: dermaPACE + Standard of care wound dressing.
- Non-energized (Inactive) Application + Standard of Care: Sham: Sham treatment (non-energized, inactive device) + Standard of care wound dressing.
- Total: Total of all reporting groups
Arm/Group | dermaPACE Application + Standard of Care | Non-energized (Inactive) Application + Standard of Care | Total
Number analyzed (Participants) | 107 | 99 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.4) | 56.2 (9.4) | 58.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 83 | 83 | 166
Region of Enrollment [Number; unit: participants]
  United States | 103 | 94 | 197
  Germany | 2 | 3 | 5
  United Kingdom | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Primary Variable for Effectiveness of the dermaPACE Device Will be Assessed by Comparing the Incidence of Complete Wound Closure of the dermaPACE and Control Groups 12 Weeks Post Initial Application.
Time Frame: 12 weeks post initial application
Population: ITT
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | dermaPACE Application + Standard of Care | Non-energized (Inactive) Application + Standard of Care
Number analyzed (Participants) | 107 | 99
participants | 22 [13.4 to 29.5] | 15 [8.7 to 23.8]

2. Secondary Outcome: Time to Wound Closure, Wound Closure Area and Volume Between Active and Control 12 Weeks Post Initial Application, Subject Pain Assessment Between Active and Control 24 Weeks Post Initial Application
Time Frame: 12 weeks post initial application and 24 weeks post initial application
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | dermaPACE Application + Standard of Care | Non-energized (Inactive) Application + Standard of Care
Serious Adverse Events (participants affected / at risk) | 34/107 | 37/99
Other Adverse Events (participants affected / at risk) | 54/107 | 42/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | dermaPACE Application + Standard of Care (N=107) | Non-energized (Inactive) Application + Standard of Care (N=99)
Application site infections (Infections and infestations) | 16 | 27
MI and cardiac failure (Cardiac disorders) | 6 | 6
GI Haemmorhage (Gastrointestinal disorders) | 2 | 2
application site disorders (General disorders) | 3 | 1
Fall, complication from other procedure (Injury, poisoning and procedural complications) | 1 | 1
bacterial test positive (Investigations) | 0 | 1
dehydration and other disease related problems (Metabolism and nutrition disorders) | 4 | 1
Arthritis and joint pain (Musculoskeletal and connective tissue disorders) | 2 | 0
ischemic attack, syncope (Nervous system disorders) | 2 | 2
renal failure (Renal and urinary disorders) | 2 | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
diabetic vascular disorder (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | dermaPACE Application + Standard of Care (N=107) | Non-energized (Inactive) Application + Standard of Care (N=99)
blood deficiencies (Blood and lymphatic system disorders) | 3 | 3
cardiac disorders (Cardiac disorders) | 4 | 1
hearing disorders (Ear and labyrinth disorders) | 4 | 1
eye conditions (Eye disorders) | 2 | 5
nausea, stomach discomfort, bowel conditions (Gastrointestinal disorders) | 12 | 16
target site pain, irritation, illnesses (General disorders) | 24 | 31
allergies (Immune system disorders) | 2 | 1
infections (Infections and infestations) | 39 | 21
non-ulcer injuries (Injury, poisoning and procedural complications) | 23 | 16
blood tests, weight increase (Investigations) | 11 | 16
anorexia, dehydration, diabetes related conditions (Metabolism and nutrition disorders) | 28 | 20
joint and muscle pain (Musculoskeletal and connective tissue disorders) | 16 | 10
skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
headache, syncope, dizziness, ischemic attack (Nervous system disorders) | 13 | 9
anxiety, depression (Psychiatric disorders) | 5 | 3
renal failure, incontinence (Renal and urinary disorders) | 3 | 6
prostatic hypoplasia, vulvovaginal burning (Reproductive system and breast disorders) | 2 | 2
coughing, congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7
blisters, dermatitis, non-ulcer skin conditions (Skin and subcutaneous tissue disorders) | 18 | 15
arterial stenosis, DVT, hypertension (Vascular disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No